CLINICAL TRIAL: NCT01717482
Title: A Pilot Study of Metformin as a Chemoprevention Agent in Non-small Cell Lung Cancer
Brief Title: Metformin as a Chemoprevention Agent in Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and funding ended
Sponsor: Mayo Clinic (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Principal Investigator, Dennis Wigle, M.D., P.h.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-006865
Record Dates: First submitted 2012-10-25; First posted 2012-10-30 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Bronchoscopy; Metformin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): Metformin 850mg twice a day
  Interventions: Drug: Metformin
- Observation (Placebo Comparator): Standard of Care Observation
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage
  Arms: Metformin
Other: Placebo Comparator — Standard of Care Observation
  Arms: Observation

SUMMARY:
The purpose of this study is to learn whether it is better to receive the drug Metformin with standard of care for lung cancer or just standard of care.

DETAILED DESCRIPTION:
Participants will need to be scheduled to undergo a surgical resection of their lung cancer at the Mayo Clinic in Rochester, Minnesota. They will be asked to provide a blood sample prior to their surgery. Samples of tumor tissue and normal lung tissue will be taken from the samples removed during your lung surgery. The tissue will be used to evaluate DNA. A skin biopsy at the edge of the incision that has already been made will be done during your surgery. We will take the skin and grow skin fibroblasts. Then we will reprogram the skin fibroblasts into induced pluripotent cells. You will be "randomized" into one of the study groups to either take Metformin for 6 months with your standard of care follow up or to receive standard of care follow up.

ELIGIBILITY:
Inclusion Criteria

* Suspected or biopsy proven Stage IA-IIIA lung squamous cell carcinoma (SCC) (must be proven SCC at the time of surgery)
* Medically fit for surgical resection (based on surgeon assessment)
* Current or prior smoker
* Age > 18 years old
* Both Male and Female
* Willing and able to consent to study, undergo study interventions, and take study drug
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Subject must start Metformin within 90 days of surgery.

Exclusion Criteria

* Currently taking metformin or other diabetic drugs
* Current or previous congestive heart failure, renal failure or liver failure
* Creatinine in Women of 1.4 or greater and Creatinine in Men of 1.5 or greater
* Existing untreated or prior cancer <5 years from diagnosis
* Received neo-adjuvant platinum-based chemotherapy or targeted therapy
* Receiving adjuvant platinum-based chemotherapy or targeted therapy after surgical resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin 850mg twice per day
  Metformin
Period: Overall Study
Arm/Group | Metformin | Observation
Started | 4 | 2
Completed | 0 | 2
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Observation | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.25 (6.87) | 62.5 (7.5) | 63 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Feasibility of Patient Randomization, Accrual, and Tissue Collection for Study Conduction
Description: To evaluate the feasibility of patient randomization, accrual, and tissue collection in a pilot study of metformin versus observation following resection of stage IA-IIIA lung squamous cell cancer for patients by assessing the reasons patients decline randomization, tracking accrual numbers, and tracking collected tissue and reasons why tissue was not collected.
Time Frame: 2 years
Population: Study terminated due to poor accrual and funding ended
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With 2-year Recurrence Free Survival
Description: To compare the 2-year recurrence free survival (RFS) rate between metformin and observation.
Time Frame: 4 years
Population: Study terminated due to poor accrual and funding ended
Groups:
- Metformin: Metformin 850mg twice a day
  Metformin
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measure Metformin Sensitivity in Induced Pluripotent Stem Cells (iPS)
Description: To develop the metformin sensitivity index based on iPS cell line metformin sensitivity measurements from the first 20 patients randomized to the metformin arm. We will then To apply the metformin sensitivity index on the remaining 25 patients randomized to metformin and the 45 observation patients (70 patients total) to compare the 2-year RFS rate between metformin-sensitive and metformin-not-sensitive patients.
Time Frame: 4 years
Population: Study terminated due to poor accrual and funding ended
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: To compare participant adverse events between metformin and observation arms using CTCAE version 4.
Time Frame: 4 years
Population: Study terminated due to poor accrual and funding ended
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a 24 months time period
Arm/Group | Metformin | Observation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=4) | Observation (N=2)
Nausea (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0)
Pleual Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stomach pain (General disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to poor accrual and funding ended

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01717482/Prot_SAP_000.pdf